CLINICAL TRIAL: NCT00779857
Title: Exclusion of the Left Atrial Appendage With the AtriClip LAA Exclusion Device in Patients Undergoing Concomitant Cardiac Surgery
Brief Title: AtriCure Exclusion of the LAA in Patients Undergoing Concomitant Cardiac Surgery
Acronym: EXCLUDE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP2008-2
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Results first posted 2013-06-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Left Atrial Appendage Exclusion
Keywords: left atrial appendage; laa; atrial fibrillation; afib; af; stroke; tia
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AtriCure LAA Exclusion System (Experimental): AtriCure LAA Exclusion System
  Interventions: Device: AtriCure LAA Exclusion System

INTERVENTIONS:
Device: AtriCure LAA Exclusion System — Exclusion of the left atrial appendage using the AtriCure LAA Exclusion System

SUMMARY:
Prospective, non-randomized trial to evaluate the safety and efficacy of the LAA Exclusion Device (Clip) for the exclusion of the LAA via epicardial tissue approximation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is greater than or equal to 18 years of age.
2. Subject has any one of the following risk factors and is thought to benefit from LAA occlusion:

   * CHADS score > 2
   * Age > 75 years
   * Hypertension and age > 65 years
   * Previous stroke
   * History of atrial fibrillation (any classification)
3. Subject is scheduled to undergo elective non-endoscopic cardiac surgical procedure(s) including cardiac surgery for one or more of the following: Mitral valve repair or replacement, Aortic valve repair or placement, Tricuspid valve repair or replacement, Coronary artery bypass procedures, concomitant surgical (ablation or cut-and-sew) Maze procedure, patent foramen ovale (PFO), atrial septal defect (ASD) repair with the device deployed while on or prepared for cardio-pulmonary bypass support.
4. Subject is willing and able to provide written informed consent.
5. Subject has a life expectancy of at least 1 year.
6. Subject is willing and able to return for scheduled follow-up visits.

Exclusion Criteria:

1. Previous cardiac surgery
2. Thrombus in the LAA/LA which cannot be evacuated prior to placement of the Clip.
3. Patients requiring surgery other than CABG and/or cardiac valve and/or surgical maze procedure and/or PFO closure and/or ASD repair.
4. NYHA Class IV heart failure symptoms
5. Need for emergent cardiac surgery (i.e. cardiogenic shock)
6. Creatinine >200 µmol/L
7. LAA is not appropriate for exclusion based on intraoperative evaluations
8. Current diagnosis of active systemic infection
9. Renal failure requiring dialysis or hepatic failure
10. A known drug and/or alcohol addiction
11. Mental impairment or other conditions which may not allow the subject to understand the nature, significance and scope of the study
12. Pregnancy or desire to get pregnant within 12-months of the study treatment
13. Preoperative need for an intra-aortic balloon pump or intravenous inotropes
14. Patients who have been treated with thoracic radiation
15. Patients in current chemotherapy
16. Patients on long term treatment with steroids not including intermittent use of inhaled steroids for respiratory diseases.
17. Patients with known connective tissue disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-09; Primary Completion 2009-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mack, MD, Principal Investigator — Baylor Heart Hospital
Locations (7):
- United States (7):
  - Macon Medical Center, Macon, Georgia
  - St. Francis Heart Hospital, Indianapolis, Indiana
  - Spectrum Health, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Carmel East Hospital, Columbus, Ohio
  - Baylor Heart Hospital, Plano, Texas
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Ailawadi G, Gerdisch MW, Harvey RL, Hooker RL, Damiano RJ Jr, Salamon T, Mack MJ. Exclusion of the left atrial appendage with a novel device: early results of a multicenter trial. J Thorac Cardiovasc Surg. 2011 Nov;142(5):1002-9, 1009.e1. doi: 10.1016/j.jtcvs.2011.07.052. Epub 2011 Sep 8. PMID 21906756

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment subjects were recruited from the routine clinical referral base of one or more surgeons at each investigational site.
Pre-assignment Details: Subjects were screened for enrollment and consented prior to being brought to the OR with the potential that they may not be eligible based on some criteria evaluated in OR (i.e. left atrial size assessed by TEE).
Groups:
- AtriCure LAA Exclusion System: AtriCure LAA Exclusion System
  AtriCure LAA Exclusion System : Exclusion of the left atrial appendage using the AtriCure LAA Exclusion System
Period: Overall Study
Arm/Group | AtriCure LAA Exclusion System
Started | 70 (70 patients treated)
30 Day Post Procedure | 68 (2 missed Visit)
3 Month Post Procedure | 65 (3 month follow-up, 65 of the subjects were available for evaluation.)
Completed | 64 (12 Month Post procedure, 64 subjects available for evaluation)
Not Completed | 6
Not completed — Death | 1
Not completed — Withdrawal by Subject | 3
Not completed — Missed Visit | 2

BASELINE CHARACTERISTICS:
Population: 70 patients treated with AtriClip LAA Exclusion System
Arm/Group | AtriCure LAA Exclusion System
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 62
Age Continuous [Mean (Standard Deviation); unit: years] | 73.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 48
Region of Enrollment [Number; unit: participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Rate of Device Related Serious Adverse Events
Description: The primary safety endpoint is the rate of device related serious adverse events within 30 days post-procedure or hospital discharge, whichever is later, compared with the rates for serious adverse events for LAA exclusion reported in the peer review literature. The safety endpoint was determined based on an independent review of all reported adverse events by an independent cardiac surgeon that was not an investigator in the study.
Time Frame: Discharge/30 days Post Procedure
Population: The primary analysis population is all patients enrolled in the trial. All available data, regardless of whether data are derived within specified time windows will be included in the analysis. Patients who do not complete the entire course of treatment will be included.
Measure: Number (95% Confidence Interval); unit: Number of participants
Arm/Group | AtriCure LAA Exclusion System
Number analyzed (Participants) | 70
Number of participants | 0 [0.00 to 0.0001]

2. Primary Outcome: Percent of Patients With Complete Occlusion of the Left Atrial Appendage.
Description: The primary efficacy endpoint is defined as the complete exclusion of the LAA defined by lack of fluid communication between the LA and LAA at both intra-operative (TEE) and 3 month (CT) evaluations and intra-operative verification of completeness of LAA exclusion.
Time Frame: 3 Months Post Procedure
Population: The primary analysis population for the efficacy endpoint is all patients enrolled into the trial who complete the intended treatment and the required post procedure and follow-up efficacy endpoint assessments (completers). All available data, regardless of whether data are derived within specified time windows, will be included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | AtriCure LAA Exclusion System
Number analyzed (Participants) | 61
percentage of subjects | 95.1 [88 to 100]

ADVERSE EVENTS:
Time Frame: Adverse events were collection from Date of Procedure through 24 month Post Procedure Follow-up.
Description: An independent Physician Adjudicator adjudicated all site reported adverse events and assessed them for seriousness and attribution to the device or the procedure. The results of the adjudication served as the basis for the summary tabulations of adverse events, including the primary safety endpoint.
Arm/Group | AtriCure LAA Exclusion System
Serious Adverse Events (participants affected / at risk) | 35/70
Other Adverse Events (participants affected / at risk) | 63/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AtriCure LAA Exclusion System (N=70)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Heparin-Induced Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (3)
Atrial Flutter (Cardiac disorders) | 2 (2)
Atrioventricular Block (Cardiac disorders) | 1 (1)
Atrioventricular Block Complete (Cardiac disorders) | 7 (7)
Bradycardia (Cardiac disorders) | 3 (3)
Cardiac Failure Congestive (Cardiac disorders) | 4 (5)
Low Cardiac Output Syndrome (Cardiac disorders) | 1 (1)
Sinoatrial Block (Cardiac disorders) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 1 (1)
Ventricular Septal Defect Acquired (Cardiac disorders) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
General Physical Health Deterioration (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1)
Bacteriaemia (Infections and infestations) | 1 (1)
Incision Site Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Drug Administration Error (Injury, poisoning and procedural complications) | 1 (1)
Drug Toxicity (Injury, poisoning and procedural complications) | 1 (1)
Operative Haemorrhage (Injury, poisoning and procedural complications) | 3 (3)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 4 (4)
Toxic Encephalopathy (Injury, poisoning and procedural complications) | 1 (1)
Traumatic Lung Injury (Injury, poisoning and procedural complications) | 1 (1)
Ejection Fraction Decreased (Investigations) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Phrenic Nerve Paralysis (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 4 (5)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic Dissection (Vascular disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 4 (4)
Hypotension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AtriCure LAA Exclusion System (N=70)
Anaemia (Blood and lymphatic system disorders) | 32 (32)
Atrial Fibrillation (Cardiac disorders) | 28 (30)
Atrioventricular Block Complete (Cardiac disorders) | 7 (7)
Bradycardia (Cardiac disorders) | 11 (11)
Cardiac Failure Congestive (Cardiac disorders) | 4 (5)
Urinary Tract Infection (Infections and infestations) | 9 (9)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (10)
Renal Failure (Renal and urinary disorders) | 7 (8)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 11 (15)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Haemorrhage (Vascular disorders) | 4 (4)
Hypotension (Vascular disorders) | 5 (5)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review communications prior to public release and can embargo communication regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the tim submitted to the sponsor for review. The sponsor can redact or modify the proposed publication to remove any language the sponsor believes would be detrimental to intellectual property or inaccurately reflect the results of the study.